CLINICAL TRIAL: NCT02539875
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2015: a Randomized Controlled Trial on Brief Intervention (AWARD Model) and Active Referral to Smoking Cessation Services
Brief Title: Promoting Smoking Cessation in the Community Via QTW 2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QTW2015
Record Dates: First submitted 2015-07-22; First posted 2015-09-03 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-11

CONDITIONS: Smoking Cessation Intervention
Keywords: Effectiveness of quit immediately (QI) and cut down to quit (CDTQ) interventions in achieving smoking abstinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AWARD, Brief leaflet, Referral leaflet, active referral (Experimental): AWARD will be delivered to smokers onsite and this includes: Ask about smoking history, Warn about the high risk, Advise to quit as soon as possible and not later than a quit date (which will qualify them for the QTW prizes), Refer smokers to smoking cessation services, and Do it again: to repeat the intervention. Brief innovative leaflet on health warning and smoking cessation. A 2-side color printed A4 leaflet will be designed to systematically cover the most important messages to motivate smoking cessation. A 2-side color printed A4 referral leaflet will be used for motivate and assist the smokers to use the smoking cessation services. the smokers will be active refer to various smoking cessation services in Hong Kong (using the referral leaflet) and motivate the smokers to use the smoking cessation services.
  Interventions: Behavioral: AWARD and brief leaflet/ Referral leaflet and active referral/ Smoking cessation booklet and general advices
- AWARD, Brief leaflet (Experimental): AWARD will be delivered to smokers onsite and this includes: Ask about smoking history, Warn about the high risk, Advise to quit as soon as possible and not later than a quit date (which will qualify them for the QTW prizes), Refer smokers to smoking cessation services, and Do it again: to repeat the intervention. Brief innovative leaflet on health warning and smoking cessation. A 2-side color printed A4 leaflet will be designed to systematically cover the most important messages to motivate smoking cessation.
  Interventions: Behavioral: AWARD and brief leaflet/ Referral leaflet and active referral/ Smoking cessation booklet and general advices
- Smoking cessation booklet, general advices (Active Comparator): Participants will receive minimal intervention, including: (1) the 12-page smoking cessation booklet (provided by COSH); (2) very brief, minimal and general smoking cessation advice include: "Please quit smoking for improving health and save money", "Please refer to the booklet for the details about smoking cessation" and "Please call us if you have any enquiry".
  Interventions: Behavioral: AWARD and brief leaflet/ Referral leaflet and active referral/ Smoking cessation booklet and general advices

INTERVENTIONS:
Behavioral: AWARD and brief leaflet/ Referral leaflet and active referral/ Smoking cessation booklet and general advices — Use AWARD and brief leaflet/ Referral leaflet and active referral/ Smoking cessation booklet and general advices interventions to achieve smoking abstinence

SUMMARY:
Although smoking prevalence is decreasing in Hong Kong, there are still 648,800 daily smokers 10.8% (Census and Statistics Department, 2013) and half will be killed by smoking (Lam, 2012) which accounts for over 7,000 deaths per year (Lam, Ho, Hedley, Mak, & Peto, 2001). Smoking also accounts for a large amount of medical cost, long-term care and productivity loss of US$688 million (0.6% Hong Kong GDP) (Census & Statistics Department, 2001; McGhee et al., 2006) . Smoking is a highly addictive behavior and it is difficult for smokers with strong nicotine dependence to quit without assistance. On the other hand, reaching and helping the many smokers who have no intention to quit is a challenge, because they are unlikely to seek professional help from smoking cessation services.

The Quit and Win programme provides an opportunity to reach and encourage a large group of smokers to make quit attempt and maintain abstinence. The Quit and Win model posits that smokers participating in the contest will have higher motivation to quit with incentives and better social support (Cahill & Perera, 2011). Studies have found that such quitting contests or incentive programs appeared to reach a large number of smokers and demonstrated a significantly higher quit rate for the quit and win group than for the control group (Cahill & Perera, 2008).

Smoking cessation services in Hong Kong are under-used with more than half (60.9%) adult daily smokers who had never used smoking cessation services (Census and Statistics Department, 2013). Among these smokers only 9.6% were willing to use the services. Existing services mostly require self-initiation to seek the services but smokers general lack the will power of initiation. Active referral will help overcome the barriers of self-initiation. There is preliminary evidence that active referral of smokers to smoking cessation hotline services may increase likelihood of smoking abstinence at 12-month follow-up compared with no active referrals (Borland et al., 2008). A recent study has also reported that individuals who used the community-based referral were also more likely to quit than those who did not (43.6% vs 15.3%, P<0.001) (Haas et al., 2015).

Therefore, the present study will examine (1) effectiveness of the active referral and AWARD approaches, (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 cigarette per day in the past 3 months
* Able to communicate in Cantonese
* Exhaled carbon monoxide (CO) 4 ppm or above, assessed by a validated CO smokerlyzer
* Have Intention to quit

Exclusion Criteria:

* Smokers who have difficulties (either physical or cognitive condition) to communicate
* Currently following other smoking cessation programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1306 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
smoking quit rate change from baseline at 3-month follow-up | 3-month follow-up
  The primary outcomes are self-reported 7-day point prevalence (pp) quit rate at 3 and 6 months among the two groups
smoking quit rate change from baseline at 6-month follow-up | 6-month follow-up
  The primary outcomes are self-reported 7-day point prevalence (pp) quit rate

SECONDARY OUTCOMES:
Biochemical validated quit rate | 3-month follow-up
  biochemically validated quit rates at 3 month in the two groups
Biochemical validated quit rate | 6-month follow-up
  biochemically validated quit rates at 6 month in the two groups
Smoking reduction rate change from baseline at 3-month follow-up | 3-month follow-up
  rate of smoking reduction by at least half of baseline amount in the two groups
Smoking reduction rate change from baseline at 6-month follow-up | 6-month follow-up
  rate of smoking reduction by at least half of baseline amount in the two groups
Smoking quit attempt change from baseline at 3-month follow-up | 3-month follow-up
  number of quit attempts at 3 month among the two groups
Smoking quit attempt change from baseline at 6-month follow-up | 6-month follow-up
  number of quit attempts at 6 month among the two groups
quit rate for all subjects change from baseline at 3-month follow-up | 3-month follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2015
Reduction rate for all subjects change from baseline at 3-month follow-up | 3-month follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2015
quit rate for all subjects change from baseline at 6-month follow-up | 6-month follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2015
Reduction rate for all subjects change from baseline at 6-month follow-up | 6-month follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2015
quit rate for all subjects change from baseline at 12-month follow-up | 12-month follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2015
Reduction rate for all subjects change from baseline at 12-month follow-up | 12-month follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2015

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Kelvin Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Council on Smoking and Health (COSH), Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Wang MP, Suen YN, Li WH, Lam CO, Wu SY, Kwong AC, Lai VW, Chan SS, Lam TH. Intervention With Brief Cessation Advice Plus Active Referral for Proactively Recruited Community Smokers: A Pragmatic Cluster Randomized Clinical Trial. JAMA Intern Med. 2017 Dec 1;177(12):1790-1797. doi: 10.1001/jamainternmed.2017.5793. PMID 29059277
- [Derived] Suen YN, Wang MP, Li WH, Kwong AC, Lai VW, Chan SS, Lam TH. Brief advice and active referral for smoking cessation services among community smokers: a study protocol for randomized controlled trial. BMC Public Health. 2016 May 11;16:387. doi: 10.1186/s12889-016-3084-z. PMID 27169630